CLINICAL TRIAL: NCT05326581
Title: Optimization of Sequences to Improve the Quality and Comfort of the Magnetic Resonance Imaging Examination
Acronym: OPTIM
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2021_30
Record Dates: First submitted 2022-03-18; First posted 2022-04-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Optimized MRI Sequences
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PATIENTS: patients benefiting from an MRI examination as part of their care
  Interventions: Device: mri
- VOLUNTEERS: healthy volunteers among staff.
  Interventions: Device: mri

INTERVENTIONS:
Device: mri — The people included will carry out an MRI comprising the sequence currently used in routine care and the different variants of the sequence being tested, for the optimization of the parameters. The duration of the examination (or the extension of the examination planned as part of patient care) will be from a few minutes to an hour depending on the sequences to be optimized. Subjects who agree to research for more than 30 minutes in the MRI machine will be compensated with a multi-brand gift voucher worth 30 euros.

SUMMARY:
The people included will carry out an MRI comprising the sequence currently used in routine care and the different variants of the sequence being tested, for the optimization of the parameters. The duration of the examination (or the extension of the examination planned as part of patient care) will be from a few minutes to an hour depending on the sequences to be optimized. Subjects who agree to research for more than 30 minutes in the MRI machine will be compensated with a multi-brand gift voucher worth 30 euros.

DETAILED DESCRIPTION:
The people included will carry out an MRI comprising the sequence currently used in routine care and the different variants of the sequence being tested, for the optimization of the parameters. The duration of the examination (or the extension of the examination planned as part of patient care) will be from a few minutes to an hour depending on the sequences to be optimized. Subjects who agree to research for more than 30 minutes in the MRI machine will be compensated with a multi-brand gift voucher worth 30 euros

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years old
* Consent to participate in the study
* Member of or beneficiary of a social security scheme
* For patients: benefiting from an MRI examination as part of their care
* For volunteers: Consent to be informed if an unexpected anomaly is revealed by the imaging.

Exclusion Criteria:

* Subject benefiting from a measure of legal protection
* Pregnant or breastfeeding women
* For volunteers: Contraindication to MRI (detailed contraindications questionnaire, THI score >28 questionnaire, hearing sensitivity questionnaire grade >1)

Min Age: 18 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participation in the study will be offered to patients performing MRI imaging as part of the treatment as well as to healthy volunteers among the staff.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Quality of imagery | Baseline
  Quality of imagery evaluated on a likert-type scale (range from : "very bad quality" to "very good quality") by two experts
Presence or absence of radiological image artifact | Baseline
  Presence/absence of radiological image artifact evaluated on a likert-type scale (range from : "major - impossible interpretation" to "none") by two experts
Confidence in diagnosis | Baseline
  Confidence in diagnosis evaluated on a likert-type scale (range from : "not confident" to "very confident") by two experts

CONTACTS AND LOCATIONS:
Overall Officials: Julien Savatovksy, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No